CLINICAL TRIAL: NCT00925119
Title: Uncoupling Protein Polymorphisms and Cardiometabolic Responses to Beta-Blockers
Brief Title: Examining Genetic Influence on Response to Beta-Blocker Medications in People With Type 2 Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Amber Beitelshees, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040291; K23HL091120 (NIH)
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Atenolol; Genetic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atenolol (Experimental): Participants will receive atenolol for 8 weeks.
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Atenolol — 12.5 mg twice daily of atenolol for 1 week; increased to 25 mg twice daily for a total of 8 weeks, if the medication is well tolerated

SUMMARY:
Beta-blockers are medications used to treat cardiovascular disease (CVD) symptoms, including high blood pressure and chest pain. People with diabetes who receive beta-blockers may experience adverse health effects, but the exact cause of why this happens remains unknown. This study will examine the genetic factors that may influence how atenolol, a beta-blocker medication, affects fat breakdown, blood sugar levels, and heart function in people with type 2 diabetes.

DETAILED DESCRIPTION:
People with diabetes who develop CVD have worse health outcomes than people without diabetes who develop CVD. Beta-blockers are medications used to treat high blood pressure, angina (i.e., chest pain), arrhythmias, and other CVD conditions. While beta-blockers are effective at treating these conditions, they may also have damaging effects on cholesterol or glucose levels, thereby possibly lessening their ability to prevent CVD events in people with diabetes. It is important to identify which patients may not benefit from receiving beta-blocker medications. Genetic factors may influence how people respond to beta-blocker medications. The purpose of this study is to evaluate the influence of genetic variation on beta-blocker-induced changes in insulin sensitivity, fat breakdown, and heart function in people with type 2 diabetes.

This study will enroll people with type 2 diabetes. At a series of up to three baseline study visits, participants will have a blood collection, a glucose tolerance test, an echocardiogram to obtain images of the heart, and biopsies of muscle from the thigh and fat from the stomach. All participants will then receive atenolol once a day for 8 weeks. During Week 1, participants will receive a low dose of atenolol. They will then attend a study visit at the end of Week 1, and study researchers will examine how well participants are tolerating the medication. If the atenolol is well tolerated, the dose will be increased. Study researchers will call participants 1 week after any dosage changes to monitor for side effects. Blood collection will occur again at a study visit at Week 4. At Week 8, participants will then attend up to three study visits for repeat baseline testing. Participants will then be slowly tapered off of atenolol over a 1-week period.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Pre-Diabetes

Exclusion Criteria:

* Insulin therapy
* Treatment with any beta-blocker in the 30 days before study entry
* Asthma
* Chronic obstructive pulmonary disease (COPD)
* Greater than first degree heart block
* Heart rate less than 60 bpm
* Systolic blood pressure less than 90 mm Hg
* Raynaud's phenomenon
* Known history of angina, heart attack, heart failure, coronary revascularization, or automatic implantable cardioverter defibrillators
* Pregnant
* Creatinine clearance less than 35 ml/min
* Hematologic dysfunction (white blood cell [WBC] count less than 3000 or hematocrit less than 28%)
* Allergy to amide anesthetics

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber L. Beitelshees, PharmD, MPH, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atenolol
Started | 31
Completed | 19
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Atenolol
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Diastolic Function (Annular Tissue Velocity [Em])
Time Frame: 8 weeks
Population: Data were not able to be collected from the echocardiography.
Arm/Group | Atenolol
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Free Fatty Acid Kinetics
Description: Estimate of peripheral lipolysis using modeling of free fatty acid levels collected during an IV glucose tolerance test. The change in threshold for insulin action (post-atenolol minus pre-atenolol) is the primary variable from this modeling that we analyzed.
Time Frame: Baseline and Week 8
Population: Modeling data not available in all subjects
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Atenolol
Number analyzed (Participants) | 5
mU/mL | 2.02 (16.5)

3. Secondary Outcome: Change in Triglycerides
Description: (Post atenolol triglycerides - Pre atenolol triglycerides)
Time Frame: Baseline and Week 8
Population: Data available in 17 subjects
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atenolol
Number analyzed (Participants) | 17
mg/dL | 17 (65)

4. Secondary Outcome: Change in Insulin Sensitivity
Description: As measured by the Homeostatic model assessment of insulin resistance (HOMA2-IR) (post atenolol - pre atenolol).
  he Homeostatic model assessment (HOMA) is a method for assessing insulin sensitivity from fasting glucose and insulin. A higher HOMA value indicates higher insulin resistance. The widely-used formulae available for HOMA1 provide only linear approximations of HOMA_%B and HOMA_IR, the inverse of HOMA_%S. These are: HOMA1_IR = [FPI (uU/ml) x FPG (mmol/l) ]/22.5 HOMA1_%B = (20 x FPI)/(FPG - 3.5) The results obtained for HOMA2 may differ considerably from HOMA1 computer-calculated values, especially for more extreme glucose and insulin values. For this reason, no attempt has been made to provide linear approximations of HOMA2 calculated values of HOMA_%B, HOMA_IR and HOMA_%S. The software needed to calculate HOMA2 values is available on this website: https://www.dtu.ox.ac.uk/homacalculator/download.php, subject to the conditions specified on the downloads page.
Time Frame: Baseline and Week 8
Population: Post and Pre atenolol data available in 17 subjects
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Atenolol
Number analyzed (Participants) | 17
arbitrary units | -0.05 (0.84)

5. Secondary Outcome: Change in Glucose Effectiveness
Description: Glucose effectiveness as measured by insulin-modified IV glucose tolerance test using the MINMOD model.
Time Frame: Baseline and Week 8
Population: Data could not be determined because assumptions for MINMOD model were not met.
Arm/Group | Atenolol
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in HDL
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atenolol
Number analyzed (Participants) | 19
mg/dL | -3.5 (5.8)

7. Secondary Outcome: Change in Insulin
Description: fasting insulin (post - pre atenolol)
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Atenolol
Number analyzed (Participants) | 17
mU/mL | -0.55 (6.03)

ADVERSE EVENTS:
Arm/Group | Atenolol
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 4/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atenolol (N=19)
Fatigue (General disorders) | 2
Bradycardia (Cardiac disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No